CLINICAL TRIAL: NCT03491917
Title: A Multi-Reader Multi-Case Controlled Clinical Trial to Evaluate the Comparative Accuracy of the Fujifilm DBT Plus S-View Versus FFDM Alone in the Detection of Breast Cancer - A Pilot Study
Brief Title: Fujifilm DBT Plus S-View Versus FFDM Alone in the Detection of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Fujifilm Medical Systems USA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FMSU2017-002A
Record Dates: First submitted 2018-01-28; First posted 2018-04-09 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- DBT plus S-View: Breast images utilizing DBT plus S-View
  Interventions: Device: DBT plus S-View
- FFDM alone: Breast images using FFDM alone only
  Interventions: Device: FFDM alone

INTERVENTIONS:
Device: DBT plus S-View — DBT plus S-View images
  Groups: DBT plus S-View
Device: FFDM alone — FFDM alone images
  Groups: FFDM alone

SUMMARY:
The purpose of this pilot is to provide credible performance estimate information in order to conduct a subsequent pivotal reader study.

DETAILED DESCRIPTION:
This clinical research is a retrospective, pilot, multi-reader, multi-case (MRMC) study with an enriched sample of 100 breast screening or diagnostic cases which were selected from the library of mammograms collected under Fujifilm protocol FMSU2013-004A (all subjects previously provided written informed consent agreeing their image data and supporting documentation could be used for future research and investigations). Approximately 6 qualified radiologists will independently perform two reads on all (approximately 100) cases. Each reader will read each case both as a FFDM (Full Field Digital Mammography) read, and a DBT (Digital Breast Tomosynthesis) plus S-View (Synthesized View) read on the ASPIRE Bellus II workstation.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects participating in FMSU2013-004A protocol with known clinical status

Exclusion Criteria:

* Female subjects that did not have known clinical status in FMSU2013-004A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This clinical research is a retrospective, pilot, multi-reader, multi-case (MRMC) study with an enriched sample of 100 breast screening or diagnostic cases which were selected from the library of mammograms collected under Fujifilm protocol FMSU2013-004A (all subjects previously provided written informed consent agreeing their image data and supporting documentation could be used for future research and investigations).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie L. Fajardo, M.D., Principal Investigator — independent contractor
Locations (1):
- International HealthCare, LLC, Norwalk, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a retrospective, multi-reader multi-case reader study. Six (6) radiologist readers read all 100 cases (half FFDM and half DBT plus S-View reads) at each of 2 visits which were separated by a memory washout period of approximately 4 weeks. Images were previously acquired under Fujifilm protocol FMSU2013-004A.
Groups:
- DBT Plus S-View; FFDM Alone: Readers will read half of the DBT plus S-View images followed by half of the FFDM only images at each of 2 sessions. There was a four week memory washout period between the 2 sessions.
Period: First Reading Session
Arm/Group | DBT Plus S-View | FFDM Alone
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0
Period: 4 Week Memory Washout Period
Arm/Group | DBT Plus S-View | FFDM Alone
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0
Period: Second Reading Session
Arm/Group | DBT Plus S-View | FFDM Alone
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DBT Plus S-View and FFDM Alone: Readers will read half of the DBT plus S-View images followed by half of the FFDM only images at each of 2 sessions. There was a four week memory washout period between the 2 sessions.
Arm/Group | DBT Plus S-View and FFDM Alone
Number analyzed (Participants) | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [51 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 91
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Compare Per Subject Average Area Under the ROC (Receiver Operating Characteristic) Curve (AUC)
Description: Compare per subject average area under the ROC curve (AUC) for DBT (Digital Breast Tomosynthesis) plus S-View (Synthesized View) versus FFDM (Full Field Digital Mammography), based on per-subject POM (probability of malignancy) scores and requiring correct lesion localization. The primary endpoint was non-inferior per-subject average AUC. Statistician estimated AUCs for each reader in each review condition (FFDM, DBT plus S-View) based on per-subject POM scores requiring correct lesion localization. Statistician also calculated for each reader the non-parametric (trapezoidal) AUC for the FFDM read, the DBT plus S-View read, and the difference between them. These AUC's, differences between them, and the associated variance-covariance matrix were obtained using the method of DeLong, et al.
Time Frame: 2 visits with 4 week washout period
Population: Retrospective images used from Fujifilm protocol FMSU2013-004A. All readers read the same 100 images in their own randomized order during 2 sessions (they read half of each modality at each session which were separated by a 4 week washout period).
Measure: Mean (95% Confidence Interval); unit: Probability
Arm/Group | DBT Plus S-View | FFDM Alone
Number analyzed (Participants) | 100 | 100
Probability | 0.819 [0.719 to 0.919] | 0.796 [0.700 to 0.891]
Statistical Analysis 1: Comparison: DBT Plus S-View vs FFDM Alone; The primary endpoint for this study was a non-inferior per-subject average area under the receiver operating characteristic (ROC) curve (AUC) requiring correct lesion localization for DBT (digital breast tomosynthesis) plus S-View (synthesized view) versus FFDM (full field digital mammography). AUCs for each reader were estimated in each review condition based on per-subject probability of malignancy (POM) scores requiring correct lesion localization; Test type: Non-Inferiority — Non-inferiority margin is delta = 0.05; p < 0.01, t-test, 2 sided — The average difference in AUC was 0.023 (two-sided 95% CI: -0.012, 0.059; non-inferiority p < 0.01 for non-inferiority margin delta = -0.05); df: 417.0 for FFDM, 424.6 for DBT plus S-View, and (1, 18.9) for the difference

ADVERSE EVENTS:
Time Frame: Approximately 5 weeks
Description: There were no AE's expected for this study, as it was a radiologist reader study utilizing retrospective imaging. No study subjects were on-site for this retrospective review. No Adverse Events to report.
Arm/Group | DBT Plus S-View | FFDM Alone
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT03491917/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT03491917/SAP_001.pdf